CLINICAL TRIAL: NCT01716351
Title: The Efficacy of Adapted Yoga in Managing Psychosocial Risk in Implantable Cardioverter Defibrillator (ICD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Stefanie Toise, Principal Investigator, Yale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #SR-1569; F31AT003757 (NIH)
Record Dates: First submitted 2012-10-17; First posted 2012-10-29 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Cardiac Arrhythmias
Keywords: Randomized Clinical Control Trial; Complementary and Alternative Medicine; Yoga; Electrophysiology; Implantable Cardioverter Defibrillator; Psychosocial; Anxiety; Self-Compassion; Anti-Tachycardia Pacing Events
MeSH Terms: conditions — Arrhythmias, Cardiac; Anxiety Disorders | interventions — Defibrillators, Implantable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adapted Yoga Intervention Group (Experimental): Patients received the Adapted Yoga Intervention for Implantable Cardioverter Defibrillator (ICD) Recipients and a call from a cardiac research nurse once monthly for five months.
  Interventions: Behavioral: Adapted Yoga Intervention for Implantable Cardioverter Defibrillator (ICD) Recipients
- Control (No Intervention): Patients received usual care and a call from a cardiac research nurse once monthly for five months to control for attention.

INTERVENTIONS:
Behavioral: Adapted Yoga Intervention for Implantable Cardioverter Defibrillator (ICD) Recipients — A weekly 80-minute standardized, repeatable adapted Yoga program designed for recipients of Implantable Cardioverter Defibrillators, including a 30-minute home practice CD.
  Arms: Adapted Yoga Intervention Group

SUMMARY:
Psychosocial risks are significant in the management of patients with cardiovascular disease and implantable cardioverter defibrillators (ICD) devices. This is a randomized, controlled, clinical study. The hypothesis is that adapted yoga (vs. usual care) will significantly reduce psychosocial risks (e.g. anxiety and depression symptoms) and improve the quality of life in ICD patients. The specialized, real-time data, collected by the device provides a unique look at the electrophysiological parameters of each patient's heart.

DETAILED DESCRIPTION:
All intervention data will be analyzed to determine the statistical significance of the data, and to accept or reject the hypothesis. In addition, the researcher will conduct supplemental interviews with patients who have lived with the implantable cardioverter defibrillator (ICD) device for at least six months and who are not in the intervention. The qualitative data gathered from these interviews will document concepts of illness and healing and general beliefs about mind-body interventions.

ELIGIBILITY:
Inclusion Criteria:

* Receipt of Implantable Cardioverter Defibrillator for 6 weeks or more
* Must be 18 or more years of age

Exclusion Criteria:

* Patients requiring more than 48 hours of hospitalization for implantation
* Mental Incompetence (Dementia)
* Physician's contra-indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-08; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Florida Shock Anxiety Scale (FSAS) | Baseline
  A 10-item list which measures patient fears about implantable cardioverter defibrillator shock.
Florida Shock Anxiety Scale (FSAS) | End of Intervention (8 weeks)
  A 10-item list which measures patient fears about implantable cardioverter defibrillator shock.
Self-Compassion Scale | Baseline
  A 26-item self-report scale that measures self-kindness, self-judgement, common humanity, isolation, mindfulness and over-identification.
Self-Compassion Scale | End of Intervention (8 weeks)
  A 26-item self-report scale that measures self-kindness, self-judgement, common humanity, isolation, mindfulness and over-identification.
The number of device-initiated ventricular defibrillations as recorded by their ICD device | Baseline
  A record of device firings from the Implantable Cardioverter Defibrillator (ICD) device data.
The number of device-initiated ventricular defibrillations as recorded by their ICD device | Six month follow-up
  A record of device firings from the Implantable Cardioverter Defibrillator (ICD) device data.
The number of anti-tachycardia pacing events among participants as recorded by their ICD device | Baseline
  As measured by each ICD device, the number of times that the device therapeutically paced the heart faster than its intrinsic rate, known as anti-tachycardia pacing (ATP), was recorded for each participant.
The number of anti-tachycardia pacing events among participants as recorded by their ICD device | End of Intervention (8 weeks)
  As measured by each ICD device, the number of times that the device therapeutically paced the heart faster than its intrinsic rate, known as anti-tachycardia pacing (ATP), was recorded for each participant.
The number of anti-tachycardia pacing events among participants as recorded by their ICD device | Six month follow-up
  As measured by each ICD device, the number of times that the device therapeutically paced the heart faster than its intrinsic rate, known as anti-tachycardia pacing (ATP), was recorded for each participant.

SECONDARY OUTCOMES:
Expression Manipulation Test | Baseline
  A 31-item list which tests personal and situational cue responsiveness.
Expression Manipulation Test | End of Intervention (8 weeks)
  A 31-item list which tests personal and situational cue responsiveness.
Pennebaker Inventory | Baseline
  A 54-item list which tests psychological responses to physical symptoms.
Pennebaker Inventory | End of Intervention (8 weeks)
  A 54-item list which tests psychological responses to physical symptoms.
State-Trait Anxiety Inventory (STAI) | Baseline
  A 30-item self report scale emphasizing dispositional states (anxiety).
State-Trait Anxiety Inventory (STAI) | End of Intervention (8 weeks)
  A 30-item self report scale emphasizing dispositional states (anxiety).
Positive Health Expectation Scale | Baseline
  A 7-item list which measures positive expectations to predict health after heart transplantation.
Positive Health Expectation Scale | End of Intervention (8 weeks)
  A 7-item list which measures positive expectations to predict health after heart transplantation.
Florida Patient Acceptance Survey (FPAS) | Baseline
  An 18-item list which measures patient acceptance of implantable cardiac device therapy.
Florida Patient Acceptance Survey (FPAS) | End of Intervention (8 weeks)
  An 18-item list which measures patient acceptance of implantable cardiac device therapy.
Center for Epidemiologic Study Depression Scale (CES-D) | Baseline
  A 20-item list which is a self-report depression scale for research in the general population.
Center for Epidemiologic Study Depression Scale (CES-D) | End of Intervention (8 weeks)
  A 20-item list which is a self-report depression scale for research in the general population.
Interpersonal Support Evaluation | Baseline
  A 16-item self-report list designed to measure belonging, self-esteem, appraisal, and other concrete areas of social support.
Interpersonal Support Evaluation | End of Intervention (8 weeks)
  A 16-item self-report list designed to measure belonging, self-esteem, appraisal, and other concrete areas of social support.
Hospitalizations | Baseline
  Medical Chart Review of cardiac and non-cardiac hospitalizations.
Hospitalizations | End of Intervention (8 weeks)
  Medical Chart Review of cardiac and non-cardiac hospitalizations.
Hospitalizations | Six month follow-up
  Medical Chart Review of cardiac and non-cardiac hospitalizations.
Implantation Status | Baseline
  Primary prevention and secondary prevention data from Medical Chart Review.
Medications | Baseline
  Review of medication use (cardiac, anti-arrhythmia, anti-depression and anti-anxiety medications) from Medical Charts.
Medications | End of Intervention (8 weeks)
  Review of medication use (cardiac, anti-arrhythmia, anti-depression and anti-anxiety medications) from Medical Charts.
Medications | Six month follow-up
  Review of medication use (cardiac, anti-arrhythmia, anti-depression and anti-anxiety medications) from Medical Charts.
Co-morbidities | Baseline
  Medical chart review for co-existing morbidities.
Co-morbidities | End of Intervention (8 weeks)
  Medical chart review for co-existing morbidities.
Co-morbidities | Six month follow-up
  Medical chart review for co-existing morbidities.
Ejection Fraction | Baseline
  Cardiac ejection fraction measured from Electro-cardiogram (EKG).
Ejection Fraction | End of Intervention (8 weeks)
  Cardiac ejection fraction measured from Electro-cardiogram (EKG).
Ejection Fraction | Six month follow-up
  Cardiac ejection fraction measured from Electro-cardiogram (EKG).
Atrial Fibrillation | Baseline
  A record of atrial events recorded in the Implantable Cardioverter Defibrillator (ICD) device data, and in Medical Chart Review.
Atrial Fibrillation | End of Intervention (8 weeks)
  A record of atrial events recorded in the Implantable Cardioverter Defibrillator (ICD) device data, and in Medical Chart Review.
Atrial Fibrillation | Six month follow up
  A record of atrial events recorded in the Implantable Cardioverter Defibrillator (ICD) device data, and in Medical Chart Review.

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie CF Toise, PhD, MPH, Principal Investigator — Yale New Haven Hospital, St. Raphael Campus; Thomas J Donohue, MD, Study Director — Yale New Haven Hospital, St. Raphael Campus